CLINICAL TRIAL: NCT01346878
Title: Antiretroviral Resistance Detection by Ultrasensitive Pyrosequencing of the HIV-1 Genome and Virological Response to Antiretroviral Rescue Treatment
Status: Completed | Type: Observational
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Other Study IDs: PRIUS-2
Record Dates: First submitted 2011-04-18; First posted 2011-05-03 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: HIV
Keywords: Ultra deep sequencing; Virological failure; Salvage antiretroviral therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to analyze the association between the baseline detection of resistance mutations through Ultra deep Sequencing (UDS) and the virological outcome of salvage antiretroviral therapy, in comparison with conventional genotypic resistance tests. Based on the data generated in this study, new resistance interpretation tools and algorithms will be developed to improve the prediction of antiretroviral therapy outcomes. The final aim of the study is to improve the clinical care of HIV-1-infected patients through the incorporation of improved new antiretroviral resistances tests in the clinical practice.

DETAILED DESCRIPTION:
Antiretroviral resistance testing is an essential tool for the clinical management of Human Immunodeficiency Virus (HIV-1)-infected persons and HIV surveillance in the community. In the absence of appropriate treatment, HIV-1 infection leads toward the collapse of the immune system and death of most HIV-1-infected persons. Adequate antiretroviral treatment usually reverses this process. Nevertheless, HIV-1 easily develops treatment resistance through the accumulation of mutations in its genome. This causes treatment failure, and the requirement of increasingly complex, toxic and expensive treatments. Resistant viruses can be transmitted to other persons. More than 10 % of HIV-1-positive persons in Spain become infected with viruses that are already resistant to at least one antiretroviral drug. Antiretroviral treatment regimens designed on the basis of drug resistance information are more efficacious, effective and efficient.

In spite of their clinical relevance, however, conventional resistance tests are insensitive and underestimate antiretroviral resistance. By means of new ultrasensitive resistance tests it is possible to detect resistant viruses in minority populations that remain undetected by conventional genotypic tests. Ultrasensitive resistance tests thus double or triple the number of patients in whom antiretroviral resistance is detected. It is important to emphasize that detection of minority resistant mutants in antiretroviral naïve patients increases more than triples the risk of virological failure. The clinical impact of detecting minority resistant variants in treatment-experienced patients with therapeutic failure remains unknown.

Recently developed techniques of parallel emulsion sequencing of thousands of amplicon clones (Ultra deep Sequencing (UDS), Roche Diagnostics/454 Life Sciences) increase the sensibility to detect polymorphisms and mutations in highly variable genomes such as in HIV-1 in several orders of magnitude. In addition, this technique allows stablishing genetic linkage of such mutations and polymorphisms in thousands of HIV-1 clonal sequences for every patient and point of follow-up. This generates an unprecedented opportunity to characterize the nature of HIV-1 variability and the physiopathology of antiretroviral resistance in depth. Ultrasensitive resistance tests hold the promise of improving the clinical management of HIV-1 seropositive patients, avoiding unnecessary toxicities, improving epidemiological estimations of antiretroviral resistance, improving the knowledge of the pathogenesis of HIV-1 infection and antiretroviral resistance, and improving the cost-efficiency of HIV-related pharmaceutical cost.

This study aims to analyze the association between the baseline detection of resistance mutations through UDS and the virological outcome of salvage antiretroviral therapy, in comparison with conventional genotypic resistance tests. Based on the data generated in this study, new resistance interpretation tools and algorithms will be developed to improve the prediction of antiretroviral therapy outcomes. The final aim of the study is to improve the clinical care of HIV-1-infected patients through the incorporation of improved new antiretroviral resistances tests in the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 18 years old, HIV +, distributed in one of the following 3 treatment groups:

   * PI GROUP: prior virologic failure of a HAART regimen including a PI (ritonavir boosted or not), and a second consecutive start HAART regimen including a PI boosted with ritonavir + 2 NRTIs. The 6 months prior to the start of the second HAART regimen, are considered as a baseline.
   * NNRTI GROUP: Virologic failure after a HAART regimen that includes 1 NNRTI and 2 NRTIs, and beginning, consecutive or not, a rescue HAART regimen with etravirine, in combination with any other drug. The 6 months before starting rescue HAART regimen with etravirine, are considered as a baseline.
   * II GROUP: Virologic failure to any prior HAART and initiation of rescue HAART including raltegravir, in combination with any other drug. The 6 months before starting rescue HAART with raltegravir are considered as a baseline.
2. Sample of 1 mL of plasma available for pyrosequencing before starting rescue HAART.
3. Viral load of HIV-1 > 5,000 copies / mL at the time of obtaining the plasma sample.
4. Any CD4 + count.
5. Availability of clinical follow-up, viral load of HIV-1 and quarterly CD4 counts to at least 48 weeks after initiation of rescue HAART.
6. Good adherence to therapy.
7. The investigation period is in any event before the start of the study.

Exclusion Criteria:

1. HIV-2 infection or HIV-1 subtype non-B.
2. Poor adherence to therapy.
3. Lack of adequate clinical and laboratory follow up.
4. Non-compliance of the patient to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * PI GROUP: prior virologic failure of a Highly active antiretroviral therapy (HAART) regimen including a Protease inhibitor (PI) (ritonavir boosted or not), and a second consecutive start HAART regimen including a PI boosted with ritonavir + 2 Nucleoside Reverse Transcriptase Inhibitor (NRTI). The 6 months prior to the start of the second HAART regimen, are considered as a baseline.
  * NNRTI GROUP: Virologic failure after a HAART regimen that includes 1 Non Nucleoside Reverse Transcriptase Inhibitor (NNRTI) and 2 NRTIs, and beginning, consecutive or not, a rescue HAART regimen with etravirine, in combination with any other drug. The 6 months before starting rescue HAART regimen with etravirine, are considered as a baseline.
  * II GROUP: Virologic failure to any prior HAART and initiation of rescue HAART including raltegravir, in combination with any other drug. The 6 months before starting rescue HAART with raltegravir are considered as a baseline.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Time to virological failure | One year

SECONDARY OUTCOMES:
Proportion of patients with VL <50 and <200 copies | week 12 and 48
Absolute decrease of viral load | week 24 and 48
Area under curve of viral load | week 24 and 48
CD4 increase | week 24 and 48
Comparison of virological failure rate associated with baseline genotypic resistance detection by conventional sequencing and ultrasensitive pyrosequencing of the HIV-1 genome. | One year
Cost-benefit analysis of minority mutant detection by ultrasensitive pyrosequencing. | Week 48

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Laboratorio de Retrovirología irsiCaixa, Badalona, Barcelona
  - Mútua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario San Cecilio, Granada, Granada
  - Hospital 12 de Octubre, Madrid, Madrid

REFERENCES:
- [Derived] Pou C, Noguera-Julian M, Perez-Alvarez S, Garcia F, Delgado R, Dalmau D, Alvarez-Tejado M, Gonzalez D, Sayada C, Chueca N, Pulido F, Ibanez L, Rodriguez C, Casadella M, Santos JR, Ruiz L, Clotet B, Paredes R. Improved prediction of salvage antiretroviral therapy outcomes using ultrasensitive HIV-1 drug resistance testing. Clin Infect Dis. 2014 Aug 15;59(4):578-88. doi: 10.1093/cid/ciu287. Epub 2014 May 29. PMID 24879788